CLINICAL TRIAL: NCT05191849
Title: Circulating Extracellular Vesicle Long RNA Profiles in the Diagnosis and Prediction of Treatment Response for Small Cell Lung Cancer
Brief Title: Circulating EV Long RNA Profiles in SCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jialei Wang, Principal Investigator, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EXRNA-SCLC-2021
Record Dates: First submitted 2021-12-23; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Small Cell Lung Cancer receiving chemotherapy (Other)
  Interventions: Diagnostic Test: Blood sample collection

INTERVENTIONS:
Diagnostic Test: Blood sample collection — Baseline blood samples are collected before chemotherapy. Dynamic blood samples are also prospectively collected after 2~4 cycles of chemotherapy, or at the time of disease progression.

SUMMARY:
To identify the circulating extracellular vesicle long RNA (exLR) profiles in small cell lung cancer (SCLC) and explore the potential of exLR as biomarkers to predict the therapeutic effect of SCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteered to participate in the study and have signed the informed consent.
2. Histological or cytological diagnosis of small cell lung cancer, and no indication of radical surgery or radiotherapy.
3. There are measurable lesions defined by RECIST standard v1.1. A lesion can be considered measurable only if the previously irradiated lesion has clear progression after radiotherapy and the previous irradiated lesion is not the sole lesion.
4. Initially treated patients who have not received any systematic therapy before. If have received postoperative adjuvant chemotherapy, the time to relapse is at least 6 months from the last adjuvant chemotherapy.
5. 18~75 years old; ECOG PS score: 0~1 points; expected survival time is more than 3 months.
6. The main organs's function meets the following criteria within 14 days before treatment:

（1）Routine blood test (without blood transfusion within 14 days): a) Hemoglobin (HB) ≥ 90 g / L; b) Absolute neutrophil (ANC) ≥ 1.5 × 109 / L; c) Platelets (PLT) ≥ 80×109/L （2）Biochemical examination: a) Total bilirubin (TBIL) ≤ 1.5 times of the upper limit of the normal (ULN); b) Alanine aminotransferase (ALT) and aspartate aminotransferase AST ≤ 2.5ULN.To patients with liver metastasis, ALT and AST ≤ 5ULN; c) Serum creatinine (Cr) ≤ 1.5ULN or creatinine clearance (CCr) ≥ 60ml / min; （3）Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ the lower limit of the normal (50%).

7. Patients with previously treated asymptomatic CNS metastases are allowed to participate in this study if all of the following criteria are met: a) No need for continuous corticosteroid therapy for CNS disease; b) No radiotherapy within 14 days prior to enrollment treatment; c) Imaging examination from the end of radiotherapy to screening period shows no CNS progression.

8. Women of childbearing age should agree to conduct contraception (such as intrauterine devices, contraceptives or condoms) during the study and within 6 months after the end of the study; and the serum or urine pregnancy test is negative within 7 days prior to study enrollment and they must be non-lactating patients; Men should agree to conduct contraception during the study and within 6 months after the end of the study.

Exclusion Criteria:

1. Histological or cytological diagnosis of small cell and non-small cell mixed lung cancer.
2. Patients who have previously received systemic chemotherapy, signal transduction inhibitors, targeted therapies, hormone and endocrine therapy.
3. Patients with other malignant tumors occurred within 5 years prior to the enrollment, except those with cured cervical carcinoma in situ and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)] , basal or squamous cell skin cancer, and localized prostate cancer and ductal breast carcinoma in situ treated with radical surgery.
4. Unresolved toxicity due to any previous treatment above CTC AE (4.0) level 2 or higher, excluding hair loss.
5. Patients with symptomatic CNS metastases.
6. Patients with uncontrolled pleural, pericardial, or peritoneal effusion requiring repeated drainage.
7. Patients with any severe and/or uncontrolled disease, including:

   1. Patients with unsatisfactory blood pressure control (systolic blood pressure >150 mmHg, diastolic blood pressure >90 mmHg).
   2. Patients with myocardial ischemia or myocardial infarction of Grade I of higher level, arrhythmia (including QTC ≥ 440ms) and congestive heart failure above Grade 2 (New York Heart Association (NYHA) classification).
   3. Patients with active or uncontrolled severe infection (≥ CTC AE Level 2).
   4. Patients with a history of immunodeficiency, including HIV-positive or other acquired, congenital immunodeficiency disease, or a history of organ transplantation.
   5. Patients with poor control of diabetes (fasting blood glucose (FBG)>10mmol/L).
   6. Patients with urine protein ≥ ++ indicated by routine urine test, and confirmed 24-hour urine protein quantitation > 1.0 g.
   7. Patients with seizures requiring treatment.
8. Patients undergone venous thrombosis events currently or within 6 months, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, and pulmonary embolism.
9. Patients with a history of psychotropic drug abuse from which they are unable to abstain or with mental disorders.
10. Patients who have participated in other clinical trials of anti-tumor drugs within four weeks.
11. Patients with severe disease that threaten the safety of themselves or affect the completion of the study according to the investigators' judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-10-25 (Estimated)

PRIMARY OUTCOMES:
Establish a model to predict curative effect | At the end of Cycle 4 (each cycle is 21 days)
  To detect the difference of exLR profiles of SCLC patients before and after treatment, and the difference of baseline exLR profiles between responders and non-responders.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China